CLINICAL TRIAL: NCT01480544
Title: Improving Maternal and Child Health in India: Evaluating Demand and Supply Side Strategies
Brief Title: Improving Maternal and Child Health in India: Evaluating Demand and Supply Side Strategies (IMATCHINE)
Acronym: IMATCHINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Stanford University (Other); International Initiative for Impact Evaluation (Other); Department for International Development, United Kingdom (Other Government); Sambodhi Research and Communication Pvt., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00031046
Record Dates: First submitted 2011-11-08; First posted 2011-11-29 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Obstetric Labor Complications; Post-partum Hemorrhage; Sepsis; Pre-eclampsia; Neonatal Mortality
Keywords: Institutional Deliveries; Maternal Health; Infant Health; Private Medical Providers; Provider Incentives; Randomized Control Trial
MeSH Terms: conditions — Obstetric Labor Complications; Postpartum Hemorrhage; Sepsis; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mothers at endline (No Intervention): Data collected on new mothers (up to three weeks after childbirth) in 180 clusters with 100 mothers in each cluster at endline.
- Treatment 1 (Experimental): Data collected on new mothers (up to three weeks after childbirth) and on providers with incentives for clinical improvements in quality of maternity care in the providers' patient populations and the catchment areas served by the providers.
  Interventions: Other: Experimental: Treatment 1
- Treatment 2 (Experimental): Data collected on new mothers (up to three weeks after childbirth) and on providers with incentives for improvement in maternal and infant health outcomes in the providers' patient populations and in the catchment areas served by the providers.
  Interventions: Other: Experimental: Treatment 2
- Control (No Intervention): Data collected on new mothers (up to three weeks after childbirth) and providers with no incentives

INTERVENTIONS:
Other: Experimental: Treatment 1 — Physicians will receive financial incentives for improving the quality of obstetric and neonatal care provided to mothers and newborns as reported by mothers during household interviews.
  Arms: Treatment 1
Other: Experimental: Treatment 2 — Physicians will receive financial incentives for improving maternal and neonatal health outcomes as reported by mothers during household interviews.
  Arms: Treatment 2

SUMMARY:
The study evaluates the impact of a new conditional cash transfer (CCT) program (Thayi Bhagya Yojana) to promote child birth in obstetric facilities in the state of Karnataka, India in order to determine its policy value and to guide efforts to improve maternal and infant health outcomes nationally. In addition, the study includes a large randomized evaluation of performance-based incentive payments to providers to improve quality of medical care provided during delivery and actual health improvement in the providers' patient populations and their catchment areas.

DETAILED DESCRIPTION:
The evaluation study will first provide new evidence on the effectiveness of demand-side strategies to increase institutional deliveries and improve childbirth outcomes. Second, the study will analyze one of the first implementations of direct rewards to providers for health improvement in a developing country. Third, the study will provide critical new insight into dynamics between demand and supply-side incentives in improving population health outcomes as either complements or substitutes.

The study uses household survey to collect data from mothers on socio-economic, human capital, quality of life variables (including below poverty line [BPL] index components) and as well as information about deliveries, fertility histories, morbidity and mortality (for mothers, infants, and children), birth related complications, health service use and spending. Additionally, provider surveys will collect data on infrastructure, staffing, provider qualifications, provider knowledge and process measures of provider performance.

ELIGIBILITY:
Inclusion Criteria:

* Households with new mothers (one to three weeks after childbirth)
* Rural private sector maternity care providers who are listed on the Karnataka government's legitimate provider list.

Exclusion Criteria:

* Households without children
* Households where mothers gave birth > 3 weeks ago
* Public sector maternity care providers
* Private sector maternity care providers serving in towns with large public providers such as Community Health Centers (CHCs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14990 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Increase institutional deliveries and improve maternal and infant health outcomes in the population. | 1 Year
  Rates of deliveries in hospitals and maternal health complications such as obstetric fistulas, post-partum hemorrhage, sepsis, as well as neonatal outcomes.

SECONDARY OUTCOMES:
Effectiveness of financial incentives to maternity care private providers for improvements in the clinical quality of services in the providers' patient populations and the catchment areas they serve. | 1 Year
  Indicators of quality of services include monitoring of the fetal heartbeat, active management of labor, and monitoring of cervical dilation and effacement.
Effectiveness of financial incentives to maternity care private providers for improvements in maternal and infant health outcomes in the providers' patient populations and the catchment areas they serve. | 1 Year
  Indicators of improvements in maternal and neonatal health outcomes include reduced incidence of maternal morbidity outcomes such as obstetric fistulas, excessive post partum bleeding, sepsis, hospital readmission, as well as neonatal outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Mohanan, PhD, MPH, Principal Investigator — Duke University
Locations (1):
- Imatchine, Bangalore, Karnataka, India